CLINICAL TRIAL: NCT01897831
Title: A Open Multi-center Clinical Study on Piperacillin Sodium and Sulbactam Sodium for Injection (2:1) for Treatment of Respiratory and Urinary Tract Infection
Brief Title: Piperacillin Sodium and Sulbactam Sodium for Injection (2:1) for Treatment of Respiratory and Urinary Tract Infection
Acronym: PIP-SBT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Xiangbei Welman Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2002 H L 0153
Record Dates: First submitted 2013-06-03; First posted 2013-07-12 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2012-09

CONDITIONS: Respiratory Tract Infections; Urinary Tract Infections
Keywords: Piperacillin Sodium and sulbactam sodium; Phase IV clinical studies; Respiratory and urinary tract infections
MeSH Terms: conditions — Respiratory Tract Infections; Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- xin te mie (Experimental): 1.5-3.0g,iv,bid or tid for 7-14 days
  Interventions: Drug: xin te mie

INTERVENTIONS:
Drug: xin te mie — durg:Piperacillin Sodium and Sulbactam Sodium for Injection(2:1) 1.5-3.0g,iv,bid for 7-14 days Serious infections:6.0-12.0g,iv,tid for 7-14 days
  Other Names: te mie jun; xin ke jun

SUMMARY:
In the proposed study, the investigators plan to evaluate the efficacy and safety of Piperacillin sodium and sulbactam sodium for injection (2:1) for the treatment of respiratory and urinary tract acute bacterial infection under the widely used in clinical conditions.

DETAILED DESCRIPTION:
Piperacillin sodium and sulbactam sodium for injection (2:1) plays a therapeutic role by the former inhibiting bacterial cell wall synthesis by irreversible competitive inhibition of β-lactamase. The antimicrobial effect of cefotaxime can be enhanced by the two combined. The compound specifically aims to the mechanism of bacterial resistance, extending the life of Piperacillin in the treatment-resistant pathogen infections.

ELIGIBILITY:
Inclusion Criteria:

1. patients who qualify for moderate and severe acute respiratory or urinary tract bacterial infection of acute bacterial infections need for systemic antibiotic therapy.
2. Age>18 years old, Gender: both
3. Women of childbearing age were to be negative pregnancy test and agree to take contraceptive measures during the trial;
4. patients were volunteers and signed informed consent form;
5. patients did not participate in other clinical trials.

Exclusion Criteria:

1. Patients were hypersusceptibility to the test drug or other penicillins ,β-lactamase inhibitor
2. Pregnant and Lactating women
3. Patients have severe liver,kidney,cardiovascular,cerebrovascular,endocrine and hematopoietic system of primary diseases and that of immunodeficiency,advanced cancer or mental illness.
4. Patients who were complicated by other diseases and thought to affect efficacy evaluations or poor compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2011-08; Primary Completion 2015-08 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
overall effect | two year
  end of treatment of bacteriological efficacy(bacterial clearance)
  The fore-and-aft changes of clinical symptoms and signs after discontinuation of drugs

SECONDARY OUTCOMES:
Number of participants with Adverse Events | two year
  the incidence(%)of allergies, skin rashes, shock,death, etc.

CONTACTS AND LOCATIONS:
Overall Officials: changqing cq li, doctor, Study Director — Chongqing Red Cross Hospital